CLINICAL TRIAL: NCT05586139
Title: Efficacy of a Food Targeting the Microbiota for a Sustained Recovery of Children With Uncomplicated Acute Malnutrition
Brief Title: Microbiome-Directed Food for Sustained Recovery From Acute Malnutrition
Acronym: MDF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government)
Collaborators: Ministry of Health, Burkina Faso (Other Government); Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Hermann Lanou, Principal Investigator, Institut de Recherche en Sciences de la Sante, Burkina Faso
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INV-016380
Record Dates: First submitted 2022-09-22; First posted 2022-10-19 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Acute Malnutrition With no Complications
MeSH Terms: interventions — milk-derived factor; S-Adenosylmethionine

STUDY DESIGN:
Intervention Model Description: Individually randomized and controlled trial,
  Stratified by severity of malnutrition:
  * 2 arms for Severe Acute malnutrition
  * 2 arms for Moderate acute Malnutrition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Microbiome-directed food (MDF) - MAM (Experimental): Each (MAM) child will receive a daily ration of MDF corresponding to his weight, for maximum 12 weeks
  Interventions: Dietary Supplement: Microbiome-directed food - MAM
- Ready-to-use supplementary food (RUSF) (Active Comparator): Each (MAM) child will receive a daily ration of MDF corresponding to his weight, for maximum 12 weeks
  Interventions: Dietary Supplement: Ready-to-use supplementary food (RUSF)
- Microbiome-directed food (MDF) - SAM (Experimental): Each (SAM) child will receive a daily ration of MDF corresponding to his weight, for maximum 12 weeks of supplementation.
  Interventions: Dietary Supplement: Microbiome-directed food (MDF) - SAM
- Ready-to-use therapeutic food (RUTF) (Active Comparator): Each (SAM) child will receive a daily ration of RUTF corresponding to his weight, for maximum 12 weeks of supplementation
  Interventions: Dietary Supplement: Ready-to-use therapeutic food (RUTF)

INTERVENTIONS:
Dietary Supplement: Microbiome-directed food - MAM — Each MAM child will be supplemented with MDF for a maximum of 12 weeks. He will be followed subsequently up to 24 weeks.
  Other Names: MDF - MAM
  Arms: Microbiome-directed food (MDF) - MAM
Dietary Supplement: Ready-to-use supplementary food (RUSF) — Each MAM child will be supplemented with RUSF for a maximum of 12 weeks. He will be followed subsequently up to 24 weeks.
  Other Names: RUSF
  Arms: Ready-to-use supplementary food (RUSF)
Dietary Supplement: Microbiome-directed food (MDF) - SAM — Each SAM child will be supplemented with MDF for a maximum of 12 weeks. He will be followed subsequently up to 24 weeks.
  Other Names: MDF - SAM
  Arms: Microbiome-directed food (MDF) - SAM
Dietary Supplement: Ready-to-use therapeutic food (RUTF) — Each SAM child will be supplemented with RUTF for a maximum of 12 weeks. He will be followed subsequently up to 24 weeks.
  Other Names: RUTF
  Arms: Ready-to-use therapeutic food (RUTF)

SUMMARY:
The goal of this experimental study is to test the efficacy of a new formulation - The microbiome-directed food (MDF) to treat acute malnutrition among children aged 6 to 23 months. The main questions are:

* Does treating children with moderate or severe uncomplicated malnutrition using MDF leads to higher programmatic recovery rate compared to standard of care ?
* Does treating children with moderate or severe uncomplicated malnutrition using MDF leads to higher sustained recovery rate compared to standard of care ? The MDF will be compared to Ready-to-use supplementary food (RUSF) for moderately malnourished children, and to Ready-to-use therapeutic food (RUTF) for severely malnourished children to see the effects on recovery and sustained recovery rate.

DETAILED DESCRIPTION:
In this stratified trial, children presenting at the health center and fulfilling the inclusion criteria will be randomly allocated into one of the study groups in a ratio of 1:1:1 for MAM and 1:1 for SAM.

The supplementation will be done on daily basis according to the child's weight for a maximum of 12 weeks, at which point the programmatic recovery assessment is done. Those who recovered before or at this point, will be subsequently followed up monthly up to 3 month for sustained recovery assessment.

Follow-up visits will be done at the health center every week for severe acute malnutrition (SAM) children and every two weeks for moderate acute malnutrition (SAM) children.

At each visit, anthropometric measurements will be performed; a morbidity questionnaire will be administered before the mother/caregiver receives the ration for the following period. For the measurement of adherence, mothers will be asked to bring back empty and unused sachets/packaging of supplements from the last visit. Questions will also be asked to the mother/caregiver on the difficulties encountered during consumption and the adverse events observed following the consumption of the supplements.

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 and 23 months
* Moderate wasting: WHZ < -2 and ≥ -3 or MUAC < 125 mm and ≥ 115mm or - Severe wasting: WHZ < -3 or MUAC < 115 mm

Exclusion Criteria:

* Bilateral pitting edema
* Not eating/lack of appetite
* Current illness medical complications requiring inpatient treatment
* Presence of any congenital abnormality or underlying chronic disease that may affect growth or risk of infection
* Known contraindication/hypersensitivity/allergy to MDCF of RUSF ingredients (chickpea flour, soy flour, banana, peanut)
* Relapse from MAM treatment or transfer from SAM treatment
* Children recently (<2 months) or enrolled in a nutrition program
* Residence outside the study area

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6200 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Programmatic recovery defined by Weight-for-height (WHZ) ≥ - 2 z-score or mid-upper arm circumference (MUAC) ≥ 125 mm | 12th weeks from admission to the supplementation program
  Moderate cute malnutrition is defined by Weight-for-height (WHZ) < - 2 z-score or mid-upper arm circumference (MUAC) < 125 mm. Higher WHZ z-score (≥ - 2) or mid-upper arm circumference (MUAC) ≥ 125 mm means better outcome synonym of recovery
Sustained recovery defined by WHZ ≥ - 2 z-score or MUAC ≥ 125 mm | 24 weeks from admission to the supplementation program
  Children who sustain recovery (WHZ ≥ - 2 z-score or MUAC ≥ 125 mm) up to 24 weeks

SECONDARY OUTCOMES:
Mean change in Weight-for-height (WHZ) z-score | 12 weeks from admission to the supplementation program
  (WHZ z-score at admission) - (WHZ z-score at 12 weeks)
Mean change in Weight-for-age (WAZ) z-score | 12 weeks from admission to the supplementation program
  (WAZ z-score at admission) - (WAZ z-score at 12 weeks)
Mean change in Height-for-age (HAZ) z-score | 12 weeks from admission to the supplementation program
  (HAZ z-score at admission) - (HAZ z-score at 12 weeks)
Time to recovery | Up to 12 weeks
  Determined by the number of days from admission to programmatic recovery among those who recovered
Dropouts | 12 weeks
  Lost to follow up
Non-response defined by WHZ < -2 z-score, or a MUAC < 125 mm | 12 weeks
  Children who failed to attain a weight-for-height (WHZ) ≥ - 2 z-score or mid-upper arm circumference (MUAC) ≥ 125 mm
Complications | up to 12 weeks
  * Edema
  * Fever >39°C or hypothermia <35°C
  * Severe dehydration
  * Repeated or incessant vomiting
  * Severe respiratory problem (IMCI criteria)
  * severe anemia (significant pallor with difficulty of breathing)
  * Severe malaria
  * Abscess or extensive skin lesions
  * Very weak, apathetic, unconscious
  * Seizure
Failure | up to 12 weeks
  Absence of weight gain, assessed at the 3rd consecutive visit;
  * Weight loss since admission to the program, assessed at the 1st visit after admission;
  * Loss of 5% of body weight compared to admission weight.

OTHER OUTCOMES:
Cost-effectiveness | 12 weeks; 24 weeks
  Cost-effectiveness, as defined by the incremental cost per child cured according to the program and per child cured sustainedly

CONTACTS AND LOCATIONS:
Overall Officials: Seni KOUANDA, MD., PhD, Principal Investigator — Institut de Recherche en Sciences de la Santé, Burkina-Faso
Locations (1):
- LANOU Hermann Bienou, Ouagadougou, Kadiogo, Burkina Faso

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lanou HB, Some JW, Koumbem MAA, Kouanda S. Microbiome-directed food to promote sustained recovery in children with uncomplicated acute malnutrition: protocol for a randomized controlled trial in Burkina Faso. BMC Nutr. 2025 May 13;11(1):92. doi: 10.1186/s40795-025-01045-x. PMID 40361242

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-07-08): https://cdn.clinicaltrials.gov/large-docs/39/NCT05586139/SAP_000.pdf